CLINICAL TRIAL: NCT07339982
Title: The Effect of Nutrient Warning vs. Traffic Light Labels and Taxation on Food Purchasing Behaviour Among UK Consumers: a Randomised Controlled Trial
Brief Title: Supermarket Labelling and Taxation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Eric Robinson, Professor Eric Robinson, University of Liverpool
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Supermarket label & tax study
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nutrition Labeling; Tax Policy
Keywords: front-of-pack labelling; nutrition labelling; traffic light label; nutrient warning label; taxation; food choice
MeSH Terms: interventions — Taxes

STUDY DESIGN:
Intervention Model Description: A 2x2 (labelling and taxation) design in which participants will be assigned to one of four conditions: (i) nutrient warning labelling and no taxation, (ii) nutrient warning labelling and taxation, (iii) current traffic light labelling and taxation or (iv) a control condition (current traffic light labelling and no taxation).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutrient warning label + no tax (Experimental)
  Interventions: Behavioral: Labelling
- Nutrient warning label + tax (Experimental)
  Interventions: Behavioral: Labelling; Behavioral: Taxation
- Traffic light label + tax (Experimental)
  Interventions: Behavioral: Labelling; Behavioral: Taxation
- Traffic light label + no tax (Active Comparator)
  Interventions: Behavioral: Labelling

INTERVENTIONS:
Behavioral: Labelling — Participants are shown food products displaying front-of pack nutrition labels (nutrient warning labels on products high in calories, saturated fat, salt, and/or sugar/traffic light labels) during a hypothetical food choice task.
Behavioral: Taxation — Food prices displayed in the hypothetical food choice task include a 20% added tax on products high in calories, saturated fat, salt, and/or sugar.
  Arms: Nutrient warning label + tax; Traffic light label + tax

SUMMARY:
Participants will be assigned to one of four conditions: (i) nutrient warning labelling and no taxation, (ii) nutrient warning labelling and taxation, (iii) current traffic light labelling and taxation or (iv) a control condition (current traffic light labelling and no taxation). Participants will complete a food ordering task using a simulated online supermarket resembling a major UK retailer (Tesco), before purchasing their selected items for delivery/collection via the retailer. Food choices will be recorded, and participants will self-report intake of purchased food items.

DETAILED DESCRIPTION:
The study will be a 2x2 (labelling and taxation) between-subjects randomised controlled trial in which participants will be recruited assigned to one of four conditions in the online survey platform "Qualtrics": (i) nutrient warning labelling and no taxation, (ii) nutrient warning labelling and taxation, (iii) current traffic light labelling and taxation or (iv) a control condition (current traffic light labelling and no taxation). In the nutrient warning labelling and no taxation condition, the corresponding warning labels will be placed on items that are high in saturated fat, salt, sugar, and/or calories. Items will be defined as 'high in' if they exceed >25% of the reference intake (RI) /100g or >30% RI/portion, consistent with the threshold for a red traffic light. RIs are established in European law (EU Regulation 1169/2011) and reflect the daily requirements of an average adult. In addition to these criteria, items will be defined as 'high in' calories if they exceed Public Health England (now UKHSA) guidelines for a meal (>600kcals/portion) or snack (>200kcals/portion). In the nutrient warning label and taxation condition, a 20% price increase (based on modelling work indicating efficacy at this level for reducing energy intake and obesity prevalence in a UK context) will also be applied to 'high in' items. In the traffic light and no taxation condition, all items will feature a traffic light label. This is broadly in line with current UK implementation (an estimated 75% of packaged products feature the label under voluntary implementation). In the traffic light label and taxation condition, a 20% price increase will also be applied to 'high in' items.

Participants will complete a food ordering task using a simulated online supermarket resembling a major UK retailer (Tesco). A subsample of items from three categories - Ready Meals for One, Starters and Sides, and Chilled Desserts - will be available for selection. All items will be from the "Tesco" brand. The subsample (8 items per category) was selected to be representative of the full sample in terms of (i) item range (i.e., cuisine type, including complementary combinations) and (ii) healthiness (i.e., similar proportions of items that are low, medium, and high across the nutrients of concern, and high/not high in energy). Ready meals that contained >1 portion, starters/sides that contained >2 portions, and desserts that contained more than >1 portion and portions that were not clearly designated (e.g., individual slices, packs) were excluded to reduce variability in item size within each category, as this could add noise to intake outcomes. The name, price, and image of the item will be displayed, consistent with the Tesco website. Item images can be clicked to display further information, such as the product description, ingredients, and nutritional information (including enlarged label), aligned with information that is presented on the Tesco website.

Participants will either be recruited via the online participant panel platform "Prolific" or via social media/a database maintained by researchers at the University of Liverpool. Participants will answer brief demographic questions, including age, sex, gender, highest education level, and annual post-tax household income (open response). Any participants completing the survey outside of Prolific will be asked to create a personal ID (first name initial, last name initial, last two digits of their phone number) which they will enter in both this survey and the follow-up survey, so that their responses can be linked. For Prolific participants, they will enter their unique Prolific ID. An attention check prompting participants to select a specific answer will be included here.

After answering demographic questions, participants will be shown instructions for the food ordering task: On the next page, a Tesco-style food selection interface will be displayed. Please choose the item(s) for yourself to be consumed for an evening meal within the next week. You are required to select one main, and can also optionally select a side, and/or a dessert. Bear in mind that you will be required to actually order, purchase, and consume these item(s).

Once participants have read the instructions, they will proceed to the Tesco-style food selection interface. Participants will be required to select one main, and, optionally, a side and/or dessert, indicated again by an on-screen "shopping list" that ticks off items as they are selected. Participants can add/remove items, navigate back-and-forth between main, side, and dessert options when making their selections, and see their selections populate a "basket" before checking out, in an interface that has been built to closely resemble the Tesco website.

After checking out, a basket summary will be displayed to participants indicating their selections. They will then be asked to open a new tab (or click the "open Tesco in a new tab" button in the survey, which opens Tesco in a new tab), and order their selected items on the Tesco website for collection/delivery within the next week. They will be told that if any of their items are unavailable, they should select what they deem to be the next-closest item available. Note - prices displayed on the Tesco website will not match those in the taxation conditions. However, we do not anticipate this to be an issue, as they will always be paying the same/less than indicated in their basket summary, and it is their initial choice that we are primarily interested in.

Participants will then be requested to upload an image/screenshot of their receipt/order confirmation, clearly indicating the items and delivery time and date. They will be asked to not include personal information (e.g., their name) in the upload. If any uploads contain personal information, this will be redacted by the researcher. They will also be asked to confirm (i) when they will receive their food (date and time) and (ii) when they will eat their food (i.e., evening of the [date]), specifying that they must adhere to this date, to aid scheduling of the follow-up survey.

After completing the ordering task, participants will answer further questions on aim guessing (open response), label and price awareness, food choice motives, representativeness of their order and the interface, and policy support. Any participants completing the survey outside of Prolific will be asked to provide their email address so that they can be contacted for the follow-up survey. Before submitting the survey, the following instructions will be displayed to participants: Thank you for answering the questions and placing your Tesco order. You will be invited to participate in a follow-up survey via [Prolific/email] the morning after you have eaten the food item(s) for your evening meal. You will receive [a reimbursement] once you have completed the follow-up survey. Please take photos of your food items before (i.e., when they are plated) and after you have finished eating, as we will ask you to upload these images in the follow-up survey. You can click the "download as PDF" button to save these instructions for your reference. Don't forget to also click the arrow to submit your survey response. If you have any questions, please contact us via [Prolific/email]. The survey will take approximately 20 minutes to complete.

The morning after participants have eaten the food items for their evening meal, they will be invited via Prolific to complete a follow-up Qualtrics survey. They will be required to upload their meal images and complete dummy questions rating each item's flavour, texture, and value for money. They will also be requested to complete a dietary recall survey for breakfast and lunch the previous day via Intake24. A unique Intake24 link will be displayed to each participant via Qualtrics based on their Prolific/personal ID number, as a clickable "open new tab" button. Participants will then return to Qualtrics to confirm their Intake24 submission Upon completion, a debrief form will automatically be displayed to participants, detailing the true study aims, sources of support, and researcher contact details. The follow-up survey will take approximately 10 minutes to complete. Any participants completing the study outside of Prolific will be asked to confirm their email address in the follow-up survey to facilitate reimbursement.

ELIGIBILITY:
Inclusion Criteria:

* Are a UK resident
* Are aged 18 years and above
* Are fluent in English
* Have access to a laptop/desktop computer with internet access
* Are willing to order, pay for, and eat a ready meal from Tesco for an evening meal
* Can access Home Delivery/Whoosh/Click & Collect from Tesco
* Do not have any major dietary restrictions (e.g., vegetarian, vegan, gluten-free)
* Are not on any medication which affects appetite
* Do not have a current or past eating disorder diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Nutritional quality of food order | Survey 1, immediately after the intervention.
  The nutritional quality of the participant's full food order will be calculated using mean-weighted UK Nutrient Profiling Model (NPM) scores (32). NPM scores are calculated by subtracting the total value of positive nutrients (fruit, vegetables & nuts, fibre, protein) from the total value of negative nutrients (calories, saturated fat, sugar, salt). Lower scores indicate better nutritional quality. To account for multiple items being selected, we will calculate a mean NPM score, weighted by the energy content of individual food items. This will be done using the 'weighted.mean' function in R (33) grouped by participant so the weights are specific to individual orders.
Likelihood of purchasing a less healthy option | Survey 1, immediately after the intervention.
  Any participants who select a less healthy item (high in at least one nutrient/energy) as part of their meal will be coded as 1, and participants who have only selected options that are not 'high in' will be coded as 0.

SECONDARY OUTCOMES:
Number of additional items purchased | Survey 1, immediately after the intervention.
  Determined based on the total number of additional items (other than the main ready meal) selected in the food choice task. Participants may choose fewer items in response to labelling/taxation.
Total energy and other nutrient intake | Survey 2, administered the morning after the Tesco order is consumed. Measured between 24 hours and one week post-intervention, depending on the scheduling of the order.
  Determined based on the total calorie, saturated fat, salt, and sugar content of all items in the Tesco order and an estimation of the proportion of each item that was consumed. Participants will take a photograph of each ordered food item before (i.e., when it is plated) and after consumption. The researcher will use the photographs to estimate the percentage consumed. Participants will also be asked whether they shared any of their meal with someone else, and if so, to estimate the percentage shared. Energy and nutrients consumed will then be calculated by multiplying the calorie/nutrient content of each item by the percentage that was consumed (considering any sharing), and adding this together across all items to calculate total energy/nutrients consumed. All percentage estimates will be independently verified by a second researcher.

OTHER OUTCOMES:
Pre-meal energy and nutrient intake | Survey 2, administered the morning after the Tesco order is consumed. Measured between 24 hours and one week post-intervention, depending on the scheduling of the order.
  In the follow-up survey, participants will complete a dietary recall questionnaire (Intake24). They will be asked to provide as much detail as possible on what they ate for breakfast and lunch on the same day that they consume their Tesco order. We anticipate that participants may compensate for their order by consuming less at prior mealtimes (or, conversely, they may consume less of their order is they consumed more at prior mealtimes). Intake24 will then produce estimates for total energy, saturated fat, salt, and sugar consumed.
Label awareness | Survey 1, immediately after the intervention.
  All participants will be asked "Did you notice any nutrition labels on the items when making your initial food choices?" (yes/no). If [yes], "What did the label(s) look like?" Response options (label name and an image of the label): Nutrient warnings, Traffic lights, NutriScore, Keyhole, Health Star Rating.
Price awareness | Survey 1, immediately after the intervention.
  All participants will be asked "Did you think about the price of the items when making your initial food choices?" (yes/no).
Policy support | Survey 1, immediately after the intervention.
  All participants will be asked (i) "If the UK Government introduced a policy that required all packaged foods high in calories, saturated fat, salt, and/or sugar to display nutrient warning labels, how would you feel?", (ii) "If the UK Government introduced a policy that required all packaged foods high in calories, saturated fat, salt, and/or sugar to be taxed so that they are 20% more expensive, how would you feel?" and (iii) "If the UK Government introduced a policy that required all packaged foods high in calories, saturated fat, salt, and/or sugar to be taxed so that they are 10% more expensive, how would you feel?" Likert scale ranging from 1-5 anchored by "Strongly oppose" and "Strongly support". The order of presentation for these questions will be randomised, and only one question will be displayed at a time.
Food choice motives | Survey 1, immediately after the intervention.
  Health and price food choice motives will be assessed using subscales from the Food Choice Questionnaire (34). The health motives subscale comprises six items (e.g., "It is important to me that the food I eat is nutritious"), while the price motives subscale contains three items (e.g., "It is important to me that the food I eat is cheap"). Items are rated on a 4-point Likert scale anchored by "Not at all important" and "Very important". Scores are then averaged within each subscale.
Representativeness of food choice and ordering interface | Survey 1, immediately after the intervention.
  "Was your food choice typical for you?" (yes/no). "Was the food choice interface typical of existing supermarket grocery ordering websites?" Likert scale ranging from 1-5 anchored by "Strongly disagree" to "Strongly agree".
Aim guessing | Survey 1, immediately after the intervention.
  Participants are initially told that the study is about evaluating supermarket ready meals. After completing the food choice task, participants will be asked what they think the real aims of the study are (open response). Any participant that guesses the study aims to be investigating the influence of food warning labels/price on food choice (or similar) will be coded as being aware of study aims. One researcher will code awareness of aims (R.E.) and a second researcher will independently verify coding.
Dummy questions | Survey 2, administered the morning after the Tesco order is consumed. Measured between 24 hours and one week post-intervention, depending on the scheduling of the order.
  In line with cover story that the study is about consumer perceptions of Tesco food products, participants will be shown three statements: "The Tesco ready meal… (i) had an enjoyable flavour, (ii) had an appealing texture and appearance, and (iii) offered good value for money". Participants will respond on a 1-5 Likert scale anchored by "Strongly disagree" and "Strongly agree".

IPD SHARING:
Plan to Share IPD: Yes
Anonymised dataset will be uploaded to the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting information will be made available upon submission of the manuscript to a journal.
Access Criteria: Any interested researchers will be able to access the anonymised dataset on the Open Science Framework.